CLINICAL TRIAL: NCT04263389
Title: Quantitative Assessment of Shoulder Proprioception in Patients With Chronic Mechanical Cervical Pain
Status: Completed | Type: Observational
Sponsor: Hamada Ahmed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Hamada Ahmed, Lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.Rec/012/002078
Record Dates: First submitted 2020-01-24; First posted 2020-02-10 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2020-02

CONDITIONS: Cervical Pain
Keywords: chronic mechanical cervical pain, shoulder proprioception,
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: control group is a normal matched group.
- study group: study group is a group of chronic mechanical cervical pain

SUMMARY:
The study was aimed to compare shoulder proprioception in chronic mechanical cervical pain to a matched normal group. This study include 2 groups, 40 subjects with mechanical chronic cervical pain and 40 healthy subjects representing the control group. The primary outcome measure was the shoulder proprioception test of both upper limbs during active repositioning and quantified with angular displacement error.

DETAILED DESCRIPTION:
The study was aimed to compare shoulder proprioception in chronic mechanical cervical pain to a matched normal group. This study include two groups, 40 subjects with mechanical chronic cervical pain and 40 healthy subjects representing the control group. The primary outcome measure was the shoulder proprioception test of both upper limbs during active repositioning and quantified with angular displacement error. Test was applied using an isokinetic dynamometer device at angle 30° for both shoulder internal and external rotation on both sides with an angular velocity 30°/sec.

ELIGIBILITY:
Inclusion Criteria:

* The age ranged from 20 to 35 years.
* Body Mass Index (BMI) between 18 and less than 30.
* Sufficient cognitive abilities that enables them to understand and follow instructions with a score more than 24 in the Mini-Mental State Examination (MMSE) scale.
* For the group with cervical pain, participants had a chronic mechanical cervical pain started from three to 12 months.
* Participants with chronic pain with a score of 3 to 65 according to the short-form of the McGill Pain Questionnaire (SF-MPQ).

Exclusion Criteria:

* Shoulder problems.
* Previous cervical or shoulder surgery.
* Shoulder or cervical trauma.
* Cervical radiculopathy.
* Sever visual and/or auditory problems.
* Cognitive impairment (a score less than 24 according to MMSE).

Ages: 20 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: For the control group they are normal subjects. For the group with cervical pain, participants had a chronic mechanical cervical pain started from three to 12 months with a score of 3 to 65 according to the short-form of the McGill Pain Questionnaire (SF-MPQ).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Absolute angular error (AAE) of shoulder joint | during the procedure
  The AAE is an angle that was measured using the isokinetic dynamometer to indicate the sense of position for shoulder joint. Two measurements were performed; AAE for external rotation range and AAE for internal rotation range for both right and left arms.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Shendy, PhD, Study Director — Associate professor Faculty of Physical Therapy-Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No